CLINICAL TRIAL: NCT01197170
Title: Hormone Receptor Positive Disease Across Solid Tumor Types: A Phase I Study of Single-Agent Hormone Blockade and Combination Approaches With Targeted Agents to Provide Synergy and Overcome Resistance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0504; NCI-2012-01794 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumors; Advanced Cancer
Keywords: Hormonal therapies; Estrogen receptor; Progesterone receptor; Hormone blockade; Hormone-positive tumors; Advanced cancer; Metastatic cancer; Avastin; Anti-VEGF monoclonal antibody; rhuMAB-VEGF; Afinitor; RAD001; Nexavar; BAY43-9006; OSI-774; Tarceva
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Anastrozole; Bevacizumab; Everolimus; Sorafenib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Anastrozole (Experimental): 1 mg PO (by mouth) daily for 28 days.
  Interventions: Drug: Anastrozole
- Anastrozole + Bevacizumab (Experimental): Anastrozole 1 mg PO daily and Bevacizumab starting dose 10 mg IV Day 1 of 21 day cycle. Expansion group added when MTD dose of Anastrozole + Bevacizumab found.
  Interventions: Drug: Anastrozole; Drug: Bevacizumab
- Anastrozole + Everolimus (Experimental): Anastrozole 1 mg PO daily and Everolimus starting dose 5 mg PO daily for 28 day cycle. Expansion group added when MTD dose of Anastrozole + Everolimus found.
  Interventions: Drug: Anastrozole; Drug: Everolimus
- Anastrozole + Sorafenib (Experimental): Anastrozole 1 mg PO daily and Sorafenib starting dose 200 mg PO twice a day for 28 day cycle. Expansion group added when MTD dose of Anastrozole + Sorafenib found.
  Interventions: Drug: Anastrozole; Drug: Sorafenib
- Anastrozole + Erlotinib (Experimental): Anastrozole 1 mg PO daily and Erlotinib starting dose 75 mg PO daily for 28 day cycle. Expansion group added when MTD dose of Anastrozole + Erlotinib found.
  Interventions: Drug: Anastrozole; Drug: Erlotinib

INTERVENTIONS:
Drug: Anastrozole — 1 mg by mouth daily of a 28 day cycle.
  Other Names: Arimidex
Drug: Bevacizumab — Starting dose 10 mg by vein on day 1 of a 21 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAB-VEGF
  Arms: Anastrozole + Bevacizumab
Drug: Everolimus — Starting dose 5 mg by mouth daily for a 28 day cycle.
  Other Names: Afinitor; RAD001
  Arms: Anastrozole + Everolimus
Drug: Sorafenib — Starting dose 200 mg by mouth twice a day of a 28 day cycle.
  Other Names: Nexavar; BAY43-9006
  Arms: Anastrozole + Sorafenib
Drug: Erlotinib — Starting dose 75 mg by mouth daily for a 28 day cycle.
  Other Names: OSI-774; Tarceva
  Arms: Anastrozole + Erlotinib

SUMMARY:
The goal of this clinical research study to find the highest tolerated dose of anastrozole alone or in combination with either everolimus (Afinitor), sorafenib (Nexavar), erlotinib (Tarceva), fulvestrant (Faslodex), or bevacizumab (Avastin) that can be given to patients with advanced cancer. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Anastrozole is designed to block the last step in estrogen (a hormone) production. In estrogen-dependent tumors, anastrozole may block tumor growth.

Sorafenib is designed to block the function of a cancer protein as well as tumor blood-vessel forming proteins. It may stop the growth of blood vessels in tumors.

Bevacizumab is designed to block or slow down the growth of cancer cells by blocking the growth of blood vessels that supply nutrients for tumor growth.

Everolimus is designed to block cancer proteins and may block tumor growth.

Erlotinib is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Fulvestrant is designed to block estrogen action. In estrogen-dependent tumors, fulvestrant may block tumor growth.

Study Drug Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group. The study staff will tell you the group you will be in.

Anastrozole Alone:

If you have not received earlier hormonal treatment, you may receive anastrozole alone.

Anastrozole Combination Groups:

If you have benefitted from hormonal treatment in the past, you may receive anastrozole combined with either bevacizumab, everolimus, sorafenib, or erlotinib.

If you are receiving treatment with a combination of drugs, you will be assigned to a dose level based on when you joined the study. Every group will receive the same dose level of anastrozole. The first group of participants will receive the lowest dose level of the second study drug (bevacizumab, everolimus, sorafenib, or erlotinib). Each new group will receive a higher dose of the second study drug than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the drug combinations are found.

Once the highest tolerated dose of the drug combinations are found, 10 extra participants will be enrolled at this dose level for each combination. This is called the expansion group.

In addition to this expansion, if a particular tumor type has responded to the study drug(s), 14 more participants with that tumor type will be enrolled at the highest safe dose level that has been found.

If your tumor starts growing again after an initial response to the combination of 2 drugs, a third drug may be added to the combination you have been taking. Depending on your current treatment one of the following drugs may be added: bevacizumab, everolimus, sorafenib, fulvestrant, or erlotinib.

Study Drug Administration:

If you take anastrozole alone or in combination with sorafenib or erlotinib or everolimus, each study "cycle" is 28 days. If you take anastrozole in combination with bevacizumab, each study "cycle" is 21 days.

You will take anastrozole by mouth 1 time every day. You can take this with or without food.

If you are assigned to take sorafenib, you will take it by mouth 1 or 2 times every day. Your doctor will tell you how often to take sorafenib. You should take sorafenib on an empty stomach either 1 hour before a meal or 2 hours after a meal.

If you are assigned to take bevacizumab, you will receive it by vein on Day 1 of every cycle. During Day 1 of Cycle 1, you will receive it over 90 minutes. The infusion time may be lowered if you tolerate the drug well.

If you are assigned to take everolimus, you will take it by mouth 1 time every day with food.

If you are assigned to take erlotinib, you will take it by mouth 1 time every day. You should take erlotinib on an empty stomach either 1 hour before eating or 2 hours after eating.

If you are assigned to receive fulvestrant, you will receive injections about one time every month. Depending on your study drug combination, you may receive 2 injections in the first month.

For the first Cycle of any of the assigned combinations you will receive the medication at MD Anderson. After the first cycle you may receive the medication with your home physician if your study doctor feels it is safe.

Study Visits:

At every visit, you will be asked if you have had any side effects.

If you take anastrozole combinations in a 28 day cycle, you will have the following tests and procedures:

During Weeks 1 and 3 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.

During Week 1 of Cycles 2 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* If your study doctor feels it is safe, you may have these follow-up visits with your home physician.

Every 3 cycles, you will have a CT scan, MRI scan, PET scan, and/or PET/CT scan to check the status of the disease. If the study doctor thinks more scans are needed, they will be performed more often.

If you take anastrozole combinations in a 21 day cycle, you will have the following tests and procedures:

During Week 1 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.

During Week 1 of Cycle 2 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* If your study doctor feels it is safe, you may have these follow-up visits with your home physician.

Every 3 cycles, you will have a CT scan, MRI scan, PET scan, and/or PET/CT scan to check the status of the disease. If the study doctor thinks more scans are needed, they will be performed more often.

Length of Study:

You may take the study drug(s) for as long as the doctor thinks it is in your best interest. You will be taken off study if you have intolerable side effects or the cancer gets worse.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

About 30 days after the last dose of study drug(s), you will have an end-of-study visit. At this visit, the following tests or procedures may be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* If the doctor thinks it is needed, you will have a CT scan, MRI scan, PET scan, and/or PET/CT to check the status of the disease.

If you have a serious side effect that lasts after the End-of-Study visit, you will be followed as long as the doctor thinks it is in your best interest.

This is an investigational study. Anastrozole, bevacizumab, everolimus, erlotinib, and sorafenib are all commercially available. Anastrozole is FDA approved to treat postmenopausal women with hormone receptor-positive early breast cancer. Bevacizumab is FDA approved to treat non-small cell lung cancer (NSCLC), colorectal cancer, breast cancer, and glioblastoma. Everolimus is FDA approved to treat advanced renal cell carcinoma. Sorafenib is FDA approved to treat advanced renal cell carcinoma, as well as hepatocellular carcinoma that cannot be removed by surgery. Erlotinib is FDA approved to treat NSCLC and pancreatic cancer. Fulvestrant is approved to treat breast cancer in postmenopausal women with estrogen receptor positive cancer.

The combination of these drugs is considered investigational.

Up to 281 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or who have had no standard therapy that induces a CR rate of at least 10% or improves survival by at least three months.
2. Measurable or non-measurable disease
3. Patients must have tumors that demonstrate ER/PR+ (positivity by IHC staining >/= 1%).
4. At least 4 weeks since the last dose of chemotherapy, immunotherapy, surgery, or radiation therapy (Exception: patients may have received palliative low dose radiation therapy one week before treatment provided it is not given to the only targeted lesions); at least 6 weeks for therapy which is known to have delayed toxicity (nitrosoureas, mitomycin-C, and liposomal doxorubicin); at least 4 weeks (or 5 half-lives, whichever is shorter) since treatment with biologic/targeted therapies; at least 2 weeks since last hormonal therapy
5. Eastern Cooperative Oncology Group (ECOG) performance status 0,1, or 2
6. Patients must have normal organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL; platelets >/= 50,000/mL; creatinine </= 2 X ULN; total bilirubin </= 2.0; ALT(SGPT) </= 3 X ULN; Exception for patients with liver metastasis: total bilirubin </= 3 x ULN; ALT(SGPT) </= 5 X ULN.
7. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
8. Ability to understand and the willingness to sign a written informed consent document
9. Female patients must either be: Post-menopausal women as defined by a. age >/= 60 years of age; b. prior bilateral oophorectomy; c. age < 60 with at least 12 months of spontaneous amenorrhea or post-menopausal range FSH and estradiol levels OR Premenopausal women receiving a gonadotropin-releasing hormone agonist.

Exclusion Criteria:

1. Patients with uncontrolled concurrent illness, including but not limited to: ongoing or active infection; altered mental status or psychiatric illness/social situations that would limit compliance with study requirements and/or obscure study results.
2. Uncontrolled systemic vascular hypertension (systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg on medication).
3. Patients with clinically significant cardiovascular disease: history of CVA within 6 months, myocardial infarction or unstable angina within 6 months, or unstable angina pectoris.
4. Women who are pregnant or breastfeeding
5. Patients with a history of bone marrow transplant within the previous two years.
6. Patients with a known hypersensitivity to any of the components of the drug products.
7. Patients unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with proper absorption of oral drugs.
8. Patients with major surgery within 30 days prior to entering the study.
9. Age under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2010-09-07 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 day cycle
  MTD defined as highest dose at which no more than 1 of 6 evaluable patients has had a dose limiting toxicity (DLT). Six patients should be treated before the dose is declared as MTD. DLTs defined as adverse events (AEs) related to study agents which occurs during the first cycle of treatment.

SECONDARY OUTCOMES:
Tumor Response | Every 21 or 28 days depending on study group
  Tumor response defined as one or more of the following: (1) stable disease for more than or equal to 4 months, (2) decrease in measurable tumor (sentinel lesions) by more than or equal to 20% by RECIST criteria, (3) decrease in tumor markers by more than or equal to 25% (for example, a ≥ 25% decrease in CA125 for patients with ovarian cancer), or (4) a partial response according to the Choi criteria, i.e. decrease in size by 10% or more, or a decrease in the tumor density, as measured in Hounsfield units (HU), by more than or equal to 15%.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wheler JJ, Moulder SL, Naing A, Janku F, Piha-Paul SA, Falchook GS, Zinner R, Tsimberidou AM, Fu S, Hong DS, Atkins JT, Yelensky R, Stephens PJ, Kurzrock R. Anastrozole and everolimus in advanced gynecologic and breast malignancies: activity and molecular alterations in the PI3K/AKT/mTOR pathway. Oncotarget. 2014 May 30;5(10):3029-38. doi: 10.18632/oncotarget.1799. PMID 24912489
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org